CLINICAL TRIAL: NCT03376191
Title: Prospective, Multicenter, Non-intervention Clinical Trial of Apatinib in the Treatment of Advanced Non-squamous，Non-small Cell Lung Cancer
Brief Title: Apatinib in Advanced Non-squamous，NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jian Fang (Other)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other); Peking University Third Hospital (Other); Peking University First Hospital (Other)
Responsible Party: Sponsor-Investigator, Jian Fang, professor, Peking University Cancer Hospital & Institute
Organization: Peking University Cancer Hospital & Institute (Other)
Other Study IDs: APTN-NIS-NSCLC-BCH
Record Dates: First submitted 2017-12-07; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Non-squamous Non-Small Cell Lung Cancer
Keywords: Apatinib; lung cancer; angiogenesis inhibitors; efficacy; safety
MeSH Terms: conditions — Lung Neoplasms | interventions — apatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: apatinib — Clinicians chose the initial dose of apatinib according to the patient's physical condition. Besides the clinicians adjusted the dose according to the patient's tolerance during the medication.The dosage was demanded not higher than 750 milligram (mg) per day. The patients received apatinib continuously, 28 days for a period, until intolerance, no longer getting benefits or patient wanted stop.

SUMMARY:
To explore the efficacy and safety of apatinib in non-squamous non-small cell lung cancer in the real-world.

DETAILED DESCRIPTION:
This is a multi-center, non-interventional clinical study. The number of patients that planned to be recruited is: from May 2017 to April 2019, the actual number of cases recruited into this study.

If the clinicians thought the patient is suitable to take apatinib treatment, and give the patient apatinib treatment, the patient can be recruited into this study. Clinicians chose the initial dose of apatinib according to the patient's physical condition. Besides the clinicians adjusted the dose according to the patient's tolerance during the medication. The dosage was demanded not higher than 750 milligram (mg) per day. The patients received apatinib continuously, 28 days for a period, until intolerance, no longer getting benefits or patient wanted stop.

During the course of the study, the researchers will not intervene the treatment of the patients, but only record the efficacy and adverse reactions.

Main evaluation criteria: PFS Secondary evaluation criteria: OS,DCR and ORR (according to RECIST1.1). Main safety indicators：AE, SAE (according to NCI CTCAE V4.0) and QOL scores (Quality of Life Questionnaire-lung cancer).

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old;
2. Histologically or cytologically confirmed, locally advanced or stage IV non-squamous, non-small cell lung cancer;
3. Regardless of the past anti-tumor treatments (no limited to the number of past treatment lines), the doctors believe that apatinib can bring benefits to patients;
4. The patient is voluntarily to join the study, and signed informed consent, good compliance, with follow-up.

Exclusion Criteria:

If any of the following criteria is met, the subject shall be excluded:

1. Squamous cell carcinoma and/or small cell lung cancer patients;
2. There are contraindications to apatinib (active bleeding, thrombosis, ulcers, intestinal perforation, intestinal obstruction, uncontrollable hypertension, grade III-IV cardiac insufficiency, major surgery within 30 days, severe liver and kidney dysfunction, etc.);
3. Allergic to apatinib and / or its excipients;
4. Pregnant or lactating women;
5. According to the researcher's judgment, there are other situations that may increase the risk associated with participating in this study or the drug, which may lead to patients not being eligible for enrollment in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Local advanced or advanced non-squamous non-small cell lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-Free survival) | From the date Into this study (signed ICF) to tumor progression or death for any reason，whichever came first, assessed up to 36 months
  From the date Into this study (signed ICF) to tumor progression or death for any reason.

SECONDARY OUTCOMES:
OS (Overall survival) | From the date Into this study (signed ICF) to death for any reason，assessed up to 60 months.
  From the date Into this study (signed ICF) to death for any reason.
DCR (Disease control rate) | From the date Into this study (signed ICF) to tumor progression，assessed up to 36 months.
  The rate of CR, PR plus SD
ORR (Objective control rate) | From the date Into this study (signed ICF) to tumor progression，assessed up to 36 months.
  The rate of CR and PR

OTHER OUTCOMES:
AE (Adverse events) | From the date Into this study (signed ICF) to 30 days after tumor progression, 30days after exit this research, or death，whichever came first, assessed up to 36 months.
  AE is classified and graded by Common Terminology Criteria for Adverse Events (CTCAE) (version 4.0).
SAE (Severe adverse events) | From the date Into this study (signed ICF) to 30 days after tumor progression, 30days after exit this research, or death，whichever came first, assessed up to 36 months.
  SAE is classified and graded by Common Terminology Criteria for Adverse Events (CTCAE) (version 4.0).
QOL scores | From the date Into this study (signed ICF) to tumor progression, exit this research, or death，whichever came first, assessed up to 36 months.
  Quality of life scores

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Didkowska J, Wojciechowska U, Manczuk M, Lobaszewski J. Lung cancer epidemiology: contemporary and future challenges worldwide. Ann Transl Med. 2016 Apr;4(8):150. doi: 10.21037/atm.2016.03.11. PMID 27195268
- [Background] Hall RD, Le TM, Haggstrom DE, Gentzler RD. Angiogenesis inhibition as a therapeutic strategy in non-small cell lung cancer (NSCLC). Transl Lung Cancer Res. 2015 Oct;4(5):515-23. doi: 10.3978/j.issn.2218-6751.2015.06.09. PMID 26629420
- [Background] Zhang H. Apatinib for molecular targeted therapy in tumor. Drug Des Devel Ther. 2015 Nov 13;9:6075-81. doi: 10.2147/DDDT.S97235. eCollection 2015. PMID 26622168
- [Background] Fontanella C, Ongaro E, Bolzonello S, Guardascione M, Fasola G, Aprile G. Clinical advances in the development of novel VEGFR2 inhibitors. Ann Transl Med. 2014 Dec;2(12):123. doi: 10.3978/j.issn.2305-5839.2014.08.14. PMID 25568876
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Background] Zhang L, Shi M, Huang C et al. A phase II, multicenter, placebo-controlled trial of apatinib in patients with advanced nonsquamous non-small cell lung cancer (NSCLC) after two previous treatment regimens. J Clin Oncol 2012; 30: Abst 7548.
- [Background] Mi YJ, Liang YJ, Huang HB, Zhao HY, Wu CP, Wang F, Tao LY, Zhang CZ, Dai CL, Tiwari AK, Ma XX, To KK, Ambudkar SV, Chen ZS, Fu LW. Apatinib (YN968D1) reverses multidrug resistance by inhibiting the efflux function of multiple ATP-binding cassette transporters. Cancer Res. 2010 Oct 15;70(20):7981-91. doi: 10.1158/0008-5472.CAN-10-0111. Epub 2010 Sep 28. PMID 20876799
- [Background] Ding L, Li QJ, You KY, Jiang ZM, Yao HR. The Use of Apatinib in Treating Nonsmall-Cell Lung Cancer: Case Report and Review of Literature. Medicine (Baltimore). 2016 May;95(20):e3598. doi: 10.1097/MD.0000000000003598. PMID 27196461
- [Background] Fan M, Zhang J, Wang Z, Wang B, Zhang Q, Zheng C, Li T, Ni C, Wu Z, Shao Z, Hu X. Phosphorylated VEGFR2 and hypertension: potential biomarkers to indicate VEGF-dependency of advanced breast cancer in anti-angiogenic therapy. Breast Cancer Res Treat. 2014 Jan;143(1):141-51. doi: 10.1007/s10549-013-2793-6. Epub 2013 Dec 1. PMID 24292957